CLINICAL TRIAL: NCT06893276
Title: Development of an eHealth Psychosocial Stress and Symptom Management Intervention for Patients With Pancreatic Cancer
Brief Title: e-Health Psychosocial Stress and Symptom Management (ePSMI) for Pancreatic Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240686; HT94252411001 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity (USARAA))
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ePSMI Group (Experimental): Participants in this group will receive the ePSMI intervention for up to ten weeks.
  Interventions: Behavioral: ePSMI

INTERVENTIONS:
Behavioral: ePSMI — Participants will complete an hour of cognitive behavioral stress management program in person or remote each week for ten weeks. The cognitive behavioral therapy (CBT) skills target reducing anxiety, (e.g., relaxation), changing negative appraisals (e.g., cognitive restructuring), coping skills training (e.g., enhancing adaptive skills), behavioral activation, interpersonal skills (e.g., communication skills) and building or enhancing social networks. The intervention will be administered online, and each module will last about 1-hour. After module completion, participants will have access to modules covered during session.

SUMMARY:
The purpose of this research is to evaluate a new, web-based program among patients with pancreatic cancer aimed at reducing psychosocial stress.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age.
2. Spanish or English speaker with ability to read one of these languages.
3. Diagnosis of pancreatic cancer.
4. Patients diagnosed with pancreatic neuroendocrine tumor (PNET).

Exclusion Criteria:

1. Patients unable to read Spanish or English, as participants will not be unable to complete surveys.
2. Have a history of severe psychiatric illness (e.g., psychosis, active suicidality, inpatient treatment in the past 12 months).
3. Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Recruited | Up to 1 year.
  Will be measured in percentages (%). The study will be considered feasible passed 60%.
Percentage of Participants Retained | Up to 1 year.
  Will be measured in percentages (%). The study will be considered feasible passed ≥ 80%.
Percentage of Study Participation | Up to 1 year.
  Will be measured in percentages (%). The study will be considered feasible passed ≥ 80%.
Number of Calls | Up to 10 weeks.
  It will be measured by number of biweekly calls.
Theoretical Framework on Acceptability Questionnaire | Up to 10 weeks.
  Scores will range from 10-50. Higher scores indicate higher acceptability.
Functional Assessment of Cancer Therapy (FACT) - Functional Hepatobiliary-Pancreatic Symptom Index (FHSI)-18 | Up to 10 weeks.
  Scores will range 0-72 with lower scores indicating better quality of life.
Patient-Reported Outcomes Measurement Information System - Pain Short Form | Up to 10 weeks.
  Scores will range 0-80 with higher scores indicating higher pain symptoms
Patient-Reported Outcomes Measurement Information System - Fatigue Short Form | Up to 10 weeks.
  Scores will range 0-80 with higher scores indicating higher fatigue symptoms
Pittsburgh Sleep Quality Index (PSQI) | Up to 10 weeks.
  Scores will range from 0-21 with higher scores indicating worse sleep quality.
Gastrointestinal Symptom Rating Scale (GSRS) | Up to 10 weeks.
  Scores will range from 0-78 with higher scores indicating worse gastrointestinal symptoms.

SECONDARY OUTCOMES:
Length of Hospital Stay | Up to 365 days.
  Measured in number of days.
Number of Participant's Readmissions | Up to 1 year.
  Measured in number of readmissions.
Number of Reoccurrence of Disease in Participants | Up to 1 year.
  Responses will be binary (yes or no). Will be measured in numbers.
Progression of Disease | Up to 1 year.
  Stages range from 0 to 4. Stage 0: carcinoma in situa Stage 1: localized Stage II: locally advanced Stage III: locally advanced with major blood vessel involvement Stage IV: Metastatic
Perceived Stress Scale | Up to 10 weeks.
  Scores will range from 0 to 40 with higher scores indicating greater perceived stress levels.
University of California, Los Angeles (UCLA) Loneliness Scale | Up tp 10 weeks.
  Scale of 20-80 with higher scores indicating higher loneliness
Interpersonal Support Evaluation List | Up tp 10 weeks.
  12 item questionnaire evaluated on a 4-point Likert scale with a higher score indicating higher support
Patient-Reported Outcomes Measurement Information System - Depression Short Form | Up to 10 weeks.
  Scores will range 0-80 with higher scores indicating higher pain symptoms
Patient-Reported Outcomes Measurement Information System - Anxiety Short Form | Up to 10 weeks.
  Scores will range 0-80 with higher scores indicating higher pain symptoms
Patient-Reported Outcomes Measurement Information System - Physical Functioning Short Form | Up to 10 weeks.
  Scores will range 0-80 with higher scores indicating higher pain symptoms
Patient-Reported Outcomes Measurement Information System - Self- Efficacy for Managing Symptoms-Short Form 8a | Up to 10 weeks.
  Scores will range 8-40 with greater scores indicating greater self- efficacy for managing symptoms.
Emotional distress measured by Measure of Current State Scale | Up to 10 weeks.
  Scores will range from 0-80 with higher scores indicating more intense emotional distress.
Difficulties in Emotional Regulation Scale | Up to 10 weeks.
  Scores will range from 18-90 with higher scores indicating less emotional regulation.
Intolerance of Uncertainty Scale | Up to 10 weeks.
  Scores will range from 27-135 with higher scores indicated greater intolerance of uncertainties.
Cancer Behavior Inventory | Up to 10 weeks.
  Scores will range from 33-297 with higher scores indicating greater self-efficacy in coping with cancer.
Emotional Bond subscale of the Multiperspective Assessment of General Change Mechanisms in Psychotherapy (MPACM-P) | Up to 10 weeks.
  Scores will range from, 5-25; higher scores indicate greater emotional connection between the therapist and patient.
Agreement of Collaboration Subscale of the Multiperspective Assessment of General Change Mechanisms in Psychotherapy (MPACM-P) | Up to 10 weeks.
  Scores will range from, 5-25; higher scores indicate greater agreement on collaboration between the therapist and patient.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Penedo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No